CLINICAL TRIAL: NCT00397059
Title: Pupillary Changes as a Potential Biomarker for Escitalopram in Relation to CYP2C19 Polymorphism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AKF-371; EudraCT no: 2006-001976-19
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Escitalopram; Pharmacokinetics; Pharmacodynamics; CYP2C19; Pupillometry; healthy volunteers
MeSH Terms: interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
To study the impact of CYP2C19 polymorphism on escitalopram pharmacokinetics and pharmacodynamics measured as changes in pupil diameter

DETAILED DESCRIPTION:
Escitalopram, the therapeutic active S-enantiomer of citalopram, is a selective serotonine reuptake inhibitor (SSRI) used for treatment of depression and anxiety disorders. The antidepressant effect is probably due to a stimulation of the serotonergic neurotransmission caused by the inhibition of the presynaptic serotonin reuptake. This inhibition may also be responsible for the increased pupil diameter seen in volunteers treated with racemic citalopram. Based on escitaloprams pharmacodynamic properties it is expected to have the same affect on pupil diameter. A dose/response relationship has not yet been established but theoretically the pupillary changes might serve as a biomarker for the serotonergic effect of escitalopram.

Escitalopram is demethylated in part by the polymorphic cytochrome P450 enzyme 2C19 (CYP2C19); but the impact of CYP2C19 polymorphism on the total metabolism of escitalopram is still to be investigated.

Objective: The aim of this study is to investigate the pharmacokinetics and pharmacodynamics in CYP2C19 extensive metabolizers (EMs) and poor metabolizers (PMs) and to investigate whether change in pupil size reaction to a light stimulus can act as a biomarker for the serotonergic effect of escitalopram.

The study will be conducted as a randomized, double blinded; placebo controlled two phases cross-over trial with single and repeated doses of 20 mg escitalopram and equivalent placebo. Sixteen healthy volunteers (8 EMs and 8 PMs) will participate in the trial. Prior to the trial, approximately 400 volunteers will be phenotyped by omeprazole metabolic ratio in order to identify the CYP2C19 EMs and PMs.

During the two phases blood samples will be drawn and pupil sizes will be measured at fixed time points after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age: 18-45 years
* Phenotyped for CYP2C19 activity

Exclusion Criteria:

* Drug or alcohol abuse
* Allergy towards escitalopram

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Dynamic pupillometry
Pharmacokinetics
AUC

SECONDARY OUTCOMES:
Cmax
Tmax
T½

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brosen, dr. med., Principal Investigator — University of Southern Denmark
Locations (1):
- Clinical Pharmacology, University of Southern Denmark, Odense, Denmark